CLINICAL TRIAL: NCT02498808
Title: Interferon-lambda: Novel Biologics for Controlling Neutrophil-mediated Pathology in Rheumatic Diseases?
Acronym: ILAND
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: Arthritis Research UK (Other)
Responsible Party: Principal Investigator, Raashid Luqmani, Professor of Rheumatology, University of Oxford
Other Study IDs: 20892
Record Dates: First submitted 2015-07-10; First posted 2015-07-15 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Arthritis; Vasculitis
Keywords: Interferon lambda; Interleukin-29; Neutrophil
MeSH Terms: conditions — Arthritis; Vasculitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Healthy controls: Staff or patients attending hospital or visitors attending with patients. They should not have vasculitis or inflammatory arthritis
- Early rheumatoid arthritis: Newly diagnosed patients with rheumatoid arthritis attending hospital, prior to use of biologic therapies
- New or relapsing ANCA vasculitis: Newly diagnosed or flaring patients with anti-neutrophil cytoplasm antibody associated systemic vasculitis attending hospital
- Newly diagnosed giant cell arteritis: Newly diagnosed patients with giant cell arteritis attending hospital

SUMMARY:
Neutrophils emerge as key immune cells in the initiation and perpetuation of immune responses in autoimmune diseases. They display marked abnormalities in phenotype and function in various autoimmune diseases, including systemic vasculitis, systemic lupus erythematosus (SLE) and rheumatoid arthritis (RA).

These neutrophils are characterised by an extended life span, increased capacity to produce reactive oxygen species, active gene expression and release of extracellular traps. Consequently, there is a need for better understanding of neutrophil phenotype and functions in these conditions, as well as for identifying molecules capable of specifically manipulating neutrophil function. The investigators have recently discovered that interferon lambdas (IFN-λs), also known as interleukin 28 (IL28) and interleukin 29 (IL29), class II cytokines with previously studied anti-viral biological functions, specifically suppress neutrophil infiltration and interleukin-1β production and thereby, halt and reverse the development of collagen induced arthritis (CIA). The investigators propose to further investigate the cellular and molecular mechanisms behind this suppression and examine the translational potential of the investigators' finding by examining the IFN-λ receptor expression and function in neutrophils isolated from the blood of healthy donors and rheumatic patients (early rheumatoid arthritis and vasculitis).

DETAILED DESCRIPTION:
Expression of Interferon lambda receptor 1 (IFNLR1)/interleukin 28 Receptor Alpha (IL28RA) in human neutrophils.

Neutrophils will be isolated from freshly drawn human blood with subsequent removal of red blood cells with dextran and/or magnetic-activated cell sorting (MACS). The investigators' preliminary results show that neutrophils isolated from the blood of a healthy donor express higher level of IL28RA messenger Ribonucleic Acid (mRNA) compared to Cluster of Differentiation-14 (CD14) negative or CD14 positive lymphocytes. To better understand the relative spread of IL28RA mRNA levels due to human heterogeneity, the investigators will compare the levels of IL28RA expression in neutrophils isolated from blood of 20 healthy donors. The investigators will examine whether treatment of human neutrophils ex vivo with recombinant human IL29 (Bristol- Meyers Squibb, BMS) induces Signal Transducer and Activators of Transcription 1 (STAT1) signalling. The investigators will also test newly generated antibodies to human IL28RA which have shown some specificity in IL28RA detection in cell lines, on neutrophil isolated from blood.

Expression of IFNLR1/IL28RA in neutrophils isolated from blood of rheumatic patients.

The investigators will then compare the levels of IL28RA expression on neutrophils isolated from blood of (1) 15 patients in the early phases of rheumatoid arthritis (RA) and while naïve to biologic therapeutic intervention; (2) 15 vasculitis patients with giant cell arteritis (GCA) (within one week of commencing high dose glucocorticoid) and (3) 15 vasculitis patients with granulomatosis with polyangitis (GPA; Wegener's) at presentation or during a relapse, prior to initiation of immunosuppressive therapy with either cyclophosphamide or rituximab. All patients will undergo standardised assessment of disease activity and damage, i.e. the Birmingham Vasculitis Activity Score version 3.0 (BVAS 3.0) and the Vasculitis Damage Index version 1.0 (VDI) for vasculitis or the disease activity score for 28 joints (DAS-28) for RA. This will allow the investigators to predict whether rheumatic patients are likely to respond to IL29 treatment.

Functional characterisation of human neutrophils treated with IL29.

The investigators will conduct a selective evaluation of the expression of adhesion molecules, the migratory responses and functional properties of human neutrophils treated with IL29 ex vivo. These selected activities will be examined in the IL29 treated neutrophils from blood of healthy donors, with or without stimulation with lipopolysaccharide (LPS), phorbol myristate acetate (PMA) or serum from RA and vasculitis patients. The investigators will assess the impact of IL29 treatment on neutrophils isolated from the blood of patients with RA and vasculitis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer or
* Recent diagnosis of rheumatoid arthritis within 1 month or
* New diagnosis of giant cell arteritis within 1 month or
* New diagnosis of anti-neutrophil cytoplasm antibody associated vasculitis within 1 month or
* Flare of anti-neutrophil cytoplasm antibody associated vasculitis within one month

Exclusion Criteria:

* Unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers will be recruited as staff or patients attending secondary care or accompanying patients but who do not have vasculitis or any form of inflammatory arthritis Patients with vasculitis or arthritis who are attending secondary care will be invited to participate if they fulfill eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Expression of IFNLR1/IL28Ra in human neutrophils, by laboratory measurement of blood neutrophils | Within one month of diagnosis (or flare of vasculitis)
  This will be tested on samples of blood taken from patients

SECONDARY OUTCOMES:
Vasculitis disease activity, based on a scale of disease activity in vasculitis (Birmingham Vasculitis Activity Score version 3.0, BVAS 3.0) | Within one month of diagnosis (or flare of vasculitis)
  This will be assessed using the patient using the Birmingham Vasculitis Activity Score (version 3.0), a questionnaire completed by the clinician. A numeric score can be calculated (range 0-63)
Vasculitis damage, based on a scale of disease damage in vasculitis (Vasculitis Damage Index version 1.0, VDI 1.0) | Within one month of diagnosis (or flare of vasculitis)
  This will be assessed using the Vasculitis Damage Index (Version 1.0), a questionnaire completed by the clinician. A numeric score can be calculated (0-64)
Disease activity assessment score for arthritis, based on a scale (Disease activity score for 28 joints, DAS-28) | Within one month of diagnosis (or flare of vasculitis)
  This will be assessed using a score of the number of painful and tender joints, results of the test of inflammatory markers (usually the C-reactive protein) and a patient's estimate of disease on a visual analogue scale. The data is recorded in a specifically designed calculator, providing a numerical score from 0 to 10
Expression of Toll like receptors, adhesion molecules and chemokine receptors in human neutrophils, by laboratory measurement of blood neutrophils | Within one month of diagnosis (or flare of vasculitis)
  This will be tested on samples of blood taken from patients.
STAT1 signalling by neutrophils | Within one month of diagnosis (or flare of vasculitis)
  This will be tested on samples of blood taken from patients.

CONTACTS AND LOCATIONS:
Overall Officials: Raashid A Luqmani, DM FRCP, Principal Investigator — Professor of Rheumatology
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, United Kingdom

REFERENCES:
- [Background] Blazek K, Eames HL, Weiss M, Byrne AJ, Perocheau D, Pease JE, Doyle S, McCann F, Williams RO, Udalova IA. IFN-lambda resolves inflammation via suppression of neutrophil infiltration and IL-1beta production. J Exp Med. 2015 Jun 1;212(6):845-53. doi: 10.1084/jem.20140995. Epub 2015 May 4. PMID 25941255
- [Background] Kotenko SV, Gallagher G, Baurin VV, Lewis-Antes A, Shen M, Shah NK, Langer JA, Sheikh F, Dickensheets H, Donnelly RP. IFN-lambdas mediate antiviral protection through a distinct class II cytokine receptor complex. Nat Immunol. 2003 Jan;4(1):69-77. doi: 10.1038/ni875. Epub 2002 Dec 16. PMID 12483210
- [Background] Sheppard P, Kindsvogel W, Xu W, Henderson K, Schlutsmeyer S, Whitmore TE, Kuestner R, Garrigues U, Birks C, Roraback J, Ostrander C, Dong D, Shin J, Presnell S, Fox B, Haldeman B, Cooper E, Taft D, Gilbert T, Grant FJ, Tackett M, Krivan W, McKnight G, Clegg C, Foster D, Klucher KM. IL-28, IL-29 and their class II cytokine receptor IL-28R. Nat Immunol. 2003 Jan;4(1):63-8. doi: 10.1038/ni873. Epub 2002 Dec 2. PMID 12469119